CLINICAL TRIAL: NCT03321383
Title: Factors Associated With Health Related Quality of Life in Patients With Functional Dyspepsia
Brief Title: Health Related Quality of Life in Functional Dyspepsia
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ari Fahrial Syam, Senior Lecture Gastroenterology Division, Principal Investigator, MD, PhD, Indonesia University
Other Study IDs: 16-08-126
Record Dates: First submitted 2017-10-18; First posted 2017-10-25 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Dyspepsia
Keywords: dyspepsia; health related quality of life
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies reported health related quality of life impairment in functional dyspepsia patients. Anxiety, depression, disease severity, age, and employment status associated with HRQOL in functional dyspepsia patients. However, data about HRQOL in Asian population was limited.This study aimed to evaluate factors associated with health related quality of life in patients with functional dyspepsia.

DETAILED DESCRIPTION:
126 functional dyspepsia patients will answer SF-36 HRQOL questionnaire, Hospital Anxiety, and Depression Scale, and Short Form Nepean Dyspepsia Index. Functional dyspepsia and Irritable Bowel Syndrome Rome III diagnostic questionnaire and GERD-Q questionnaire will be used to determine FD type and IBS or GERD overlap.

ELIGIBILITY:
Inclusion Criteria:

* Dyspepsia patients
* Normal or non ulcer esophagogastroduodenescopy finding

Exclusion Criteria:

* History of GI bleeding
* History of GI malignancies
* Hepatobiliary tract disease
* Diabetes mellitus
* Chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Functional dyspepsia patients at Gastroenterology Clinic in Cipto Mangunkusumo Hospital Jakarta
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | 1 month
  Short Form -36 health survey includes one scale for each of eight measured health domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. These eight domains aggregates into physical component summary and mental component summary. All health domain scales are scored using norm-based scores ranging 0 to 100 with higher scores indicate better health

SECONDARY OUTCOMES:
Anxiety | 2 weeks
  The Hospital anxiety and depression scale (Anxiety score) This consists of seven questions on anxiety on 4 point (0-3) response category. Total score range 0-21.
Depression | 2 weeks
  The Hospital anxiety and depression scale (Depression score). This consists of seven questions on depression on 4 point (0-3) response category. Total score range 0-21.
Dyspepsia symptoms severity | 2 weeks
  Nepean dyspepsia index (NDI) score. 10-item questionnaire measuring symptoms and health-related quality of life in functional dyspepsia. Each item is measured on a 5 point Likert Scale ranging from 0 (not at all) to 4 (extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Ari F Syam, MD, PhD, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hantoro IF, Syam AF, Mudjaddid E, Setiati S, Abdullah M. Factors associated with health-related quality of life in patients with functional dyspepsia. Health Qual Life Outcomes. 2018 May 2;16(1):83. doi: 10.1186/s12955-018-0913-z. PMID 29720190